CLINICAL TRIAL: NCT01260116
Title: Efficacy and Safety of Ziprasidone in the Treatment of Depressive Symptoms in Patients With Schizophrenia：an 8-week Open-label Study
Brief Title: Efficacy and Safety of Ziprasidone to Treat Depressive Symptoms in Patients With Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wuhan University (Other)
Collaborators: Peking University (Other); Pfizer (Industry)
Responsible Party: Weidong Xiao, Renmin hospital of Wuhan University
Other Study IDs: WS897429
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: The Primary Evaluation is the Change From Baseline at End of Study for CDSS Total Scores.; The Secondary Efficacy Evaluations Include: MADRS, PANSS Total Scores and Subscales and Responder Rate; CGI-S and CGI-I Scales.; Safety Evaluations Include: Laboratory Test Abnormalities; BARS and SAS; Physical Examinations; Vital Signs; Electrocardiogram,Etc.; Subjective Well-being Under Neuroleptics Short Form Will be Used in Our Study to Assess the Subjective Side-effects.
Keywords: Efficacy,safety,ziprasidone,depressive symptoms ,schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Ziprasidone,Zeldox capsule

SUMMARY:
This study is going to determine the efficacy, tolerability and safety of ziprasidone in 120 schizophrenic patients with depressive symptoms. The study will be carried out at 2 mental centers in China. Subjects will be required to attend the center at screening, baseline, Weeks 1, 2, 4 ,6 and 8 or early termination visit.

At screening, patients underwent psychiatric and physical examination, standard lab tests, and an Electrocardiograph.

At baseline, if they continued to be eligible, they began ziprasidone 20 mg twice daily.

Depending on response and tolerability, ziprasidone could be gradually escalated to a maximum of 80 mg twice daily.

DETAILED DESCRIPTION:
Primary objective The primary objective was to evaluate the efficacy of ziprasidone in the treatment of depressive symptoms in patients with schizophrenia.

Secondary objectives The secondary objective was to evaluate the efficacy and the safety and tolerability of ziprasidone in the treatment of schizophrenic patients with depressive symptoms.

Study design This study was going to determine the efficacy, tolerability and safety of ziprasidone in 120 schizophrenic patients with depressive symptoms. The study was carried out at 2 mental centers in China. Subjects were required to attend the center at screening, baseline, Weeks 1, 2, 4 ,6 and 8 or early termination visit.

At screening, patients underwent psychiatric and physical examination, standard lab tests, and an Electrocardiograph.

At baseline, if they continued to be eligible, they began ziprasidone 20 mg twice daily.

Depending on response and tolerability, ziprasidone could be gradually escalated to a maximum of 80 mg twice daily.

Dosage/Administration

At baseline subjects received study drug according to the following regimen:

Day 1-2: ziprasidone 20 mg twice daily. Day 3-4: ziprasidone 40 mg twice daily. Day 5-6: ziprasidone 60 mg twice daily. Day 7-Week 8: ziprasidone 40, 60 or 80 mg twice daily. At visit 3 (week 1) the dosage of study drug was titrated up or down based on the clinical status of the subject and the safety and tolerability of the study drug. Subjects received all study drugs with food and under supervision.

Treatment Duration It's a 8 weeks' study. There are 7 visits in this study. Visit 1 is screening visit; Visit 2 is baseline visit; Visit 3 is Week 1; Visit 4 is Week 2; Visit 5 is Week 4; Visit 6 is Week 6; Visit 7 is Week 8.

ELIGIBILITY:
Inclusion Criteria:

* (1).First-episode or non-refractory recurrent male or female in-hospitalized subjects (aged 18 to 65 years) with a diagnosis of schizophrenia and a minimum score of 70 on the Positive and Negative Syndrome Scale (PANSS) at randomization. First-episode is defined as duration of illness from the onset of psychotic symptoms ranged from 3 days to 36 months and without systemic treatment. Refractory is defined as failure to experience a therapeutic response during acute exacerbation following adequate trials of marketed antipsychotic agents on two or more occasions during the two years prior to study entry.

  (2).Patients who meet DSM-IV-TR criteria for schizophrenia and have been diagnosed as having "295.XX schizophrenia".

  (3).Patients with a CDSS total score of 5 or more in screening visit and baseline visit.

  (4).Patients or their guardian have the ability to understand and to provide informed consent to the examination, observation, and evaluation processes specified in this protocol, and have signed the informed consent from based on a full understanding of the trial.

Exclusion Criteria:

* (1).Patients who have received systemic treatment of any antipsychotics or antidepressants within 12 weeks prior to informed consent.

  (2).Women who are pregnant, possibly pregnant, or breast-feeding. (3).Patients with psychotic symptoms that are clearly due to another general medical condition or direct physiological effects of a substance.

  (4).Patients who have met DSM-IV-TR criteria for a substance-related disorder within 3 months (90 days) prior to informed consent (excluding caffeine- and nicotine-related disorders but including abuse of benzodiazepines) (5).Patients who have received ECT treatment within 8 weeks prior to informed Consent.

  (6).Patients who have used supplements containing centrally-acting substances (tryptophan, St. John's wort) within 4 weeks prior to informed consent.

  (7).Patients with unstable thyroid disorder (hypothyroidism, hyperthyroidism) or those who have received thyroid treatment within 3 months (90 days) prior to informed consent.

  (8).Patients considered to be unresponsive to clozapine (9).Patients at significant risk of developing a severe adverse event. Patients who have a medical condition that would interfere with assessments of safety or efficacy during the course of the study, or who have a history of such a condition. For example, patients diagnosed as having a complication of serious hepatic, renal, cardiac, or hematopoietic disorder, such as those described below, within 4 weeks prior to informed consent or during the screening period Hepatic disorder: Total bilirubin≥3.0 mg/dL, AST (GOT) and ALT(GPT)≥2.5 times the upper limits of normal levels Renal disorder: Creatinine ≥ 2 mg/dL Cardiac disorder: patients with a known history of QT prolongation (including congenital long QT syndrome); patients with recent acute myocardial infarction; patients with uncompensated heart failure (10).Patients known to have a history or complication of allergy to ziprasidone or other quinolinone-skeleton compounds (11).Patients with a history or a complication of neuroleptic malignant syndrome (12).Patients who represent a significant risk of committing suicide (13).Patients with a history or a complication of organic brain disorder or convulsive disorder, such as epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First-episode or non-refractory recurrent male or female in-hospitalized subjects (aged 18 to 65 years) with a diagnosis of schizophrenia company with depressive symptoms
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-10 (Estimated); Study Completion 2012-03 (Estimated)